CLINICAL TRIAL: NCT06908889
Title: Characterization of Bacterial and Mycosis Skin Flora in Seborrheic Macular Hypopigmentation - Microbiome_SHM
Brief Title: Characterization of Bacterial and Mycosis Skin Flora in Seborrheic Macular Hypopigmentation - Microbiome
Acronym: Microbiome_SHM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 24-PP-17
Record Dates: First submitted 2025-03-17; First posted 2025-04-03 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Hypopigmentation
MeSH Terms: conditions — Hypopigmentation

STUDY DESIGN:
Intervention Model Description: The study schedule consists of two on-site visit (inclusion and followup). Skin swabs will be obtained from the patient's facial lesional (FLS) and perilesional sites (FPS) located in the same facial area but at least 1 cm away from any hypopigmented macules. One skin swab will be obtained in healthy volunteers matched on sex, age, skin type and location of the skin sample.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients (Other): The study population will consist of adult subjects (≥ 18 years) with Seborrheic Macular Hypopigmentation.
  Interventions: Other: Skin's lesion patients
- Vulunteers (Other): Volunteers will be included once the required number of SMP patients has been attained. Volunteers are going to be recruited only at the coordinator center, the CHU of Nice. Recruitment will be communicated to medical and/or Inserm staff, via an announcement in the respective departments.
  Interventions: Other: Skin's lesion vulunteers

INTERVENTIONS:
Other: Skin's lesion patients — Skin swabs will be obtained from the patient's facial lesional (FLS) and perilesional sites (FPS) using a sterile cotton swab. The microbiota of the same anatomical face regions will be collected on volunteers, once the 10 SMH patients have been enrolled. The swab is premoistened in a specific cocktail solution and rubbed onto the skin surface for 45sec. The pressure during the sampling involves rubbing the area of interest with a smear over the entire zone. The skin reddens slightly under the exerted pressure.
  Arms: Patients
Other: Skin's lesion vulunteers — Skin swabs will be obtained from the patient's facial lesional (FLS) and perilesional sites (FPS) using a sterile cotton swab. The microbiota of the same anatomical face regions will be collected on volunteers, once the 10 SMH patients have been enrolled. The swab is premoistened in a specific cocktail solution and rubbed onto the skin surface for 45sec. The pressure during the sampling involves rubbing the area of interest with a smear over the entire zone. The skin reddens slightly under the exerted pressure.
  Arms: Vulunteers

SUMMARY:
Hypopigmented skin changes are commonly encountered by dermatologists. A new dermatological entity was identified as scattered, hypopigmented oval-shaped macules and patches distributed mostly in seborrheic area of the face and of the trunk in dark skinned individuals. This patterned presentation of hypopigmentation was first described in the literature under the name of hypochromic vitiligo or vitiligo minor. Nerveless, histopathological patient's specimens analyzed by Krueger et al. clearly highlight that there is no tangible causal correlation with a diagnosis of vitiligo. They propose to rename this entity to Seborrheic Macular Hypopigmentation (SMH). The etiopathology of this dermatosis is still unknown preventing to propose any satisfactory treatment for this disfiguring affection.The objective of this study is to analyze the bacterial and fungal skin microbiome on hypochromic lesions of SMH compared to the surrounding non-lesional skin of the same patients and to healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Female and male patients ≥ 18 years of age
2. Clinical diagnosis of SMH with lesion of the face
3. Written informed consent obtained before any assessment is performed
4. Affiliation with a social security scheme
5. Physical and psychological ability to participate

Exclusion Criteria:

1. Use of systemic antibiotics or any systemic antifungal treatments within 4 weeks before the inclusion visit
2. Use of topical antibiotics or any topical antifungal treatments on the face within 2 weeks before the inclusion visit
3. Use of any topical cream, gel, serum or ointment within 2 days before the inclusion visit
4. Laser, radiofrequency, peeling or any other procedure on the face in the past 3 months before the inclusion visit
5. Vulnerable patients: minors, patients under guardianship or curatorship, pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2026-01-25 (Estimated); Study Completion 2026-06-25 (Estimated)

PRIMARY OUTCOMES:
The bacterial skin microbiome of SMH patients vs voluntheers | at baseline
  For each sample, the bacterial profiles determined by real time PCR, will be described and compared as follows: seborrheic macular hypopigmented lesions versus same anatomic area in healthy volunteers.

SECONDARY OUTCOMES:
The bacterial skin microbiome of SMH patients compare to the non-lesional surrounded skin of the same patients. | at baseline
  For each sample, the bacterial profiles determined by real time PCR, will be described and compared as follows: intra-individual hypochromic macula lesions versus perilesional areas located at least 1cm away from any hypopigmented macules.

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Passeron, PhD, Principal Investigator — CHU de Nice, Service de Dermatologie
Locations (3):
- France (3):
  - CHU de Nice - Hôpital de l'Archet, Nice, Alpes-Maritimes
  - Hôpital Louis Pasteur, hôpitaux Civils de Colmar, Colmar, Colmar
  - Hôpital Saint-Louis - APHP, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No